CLINICAL TRIAL: NCT02985164
Title: Radiation Exposure Affecting Anaesthesia Personnel During Endoscopic Retrograde Cholangiopancreatography
Brief Title: Radiation Exposure During Endoscopic Retrograde Cholangiopancreatography
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Siriraj Hospital (Other)
Responsible Party: Principal Investigator, Phawan Suton, Nurse Anesthetist, Siriraj Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 270/2558(EC2)
Record Dates: First submitted 2016-11-27; First posted 2016-12-07 (Estimated); Last update posted 2016-12-07 (Estimated); Status verified 2016-12

CONDITIONS: Cholangiopancreatography, Endoscopic Retrograde; Occupational Exposure; Radiation Injuries
Keywords: Anesthesiology( H02.403.066 ); Radiation Protection( N06.850.810.425); Cholangiopancreatography, Endoscopic Retrograde(D002760 )
MeSH Terms: conditions — Radiation Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PDSa (Pocket radiation dosimeter a) (Experimental): A co-researcher reset and prepared 4 pocket dosimeters (PDS) and labelled as PDSa1, PDSa2, PDSb1 and PDSb2.
  The PDSa1 and PDSa2 were placed on the outside and inside of a lead shirt respectively. The shirt-covered box was close to an anesthetic machine. This box would represent anesthetic personnel on duty and marked as position A. Position A was 160 cm. above the floor
  Interventions: Radiation: PDSa
- PDSb (Pocket radiation dosimeter b) (Experimental): The PDSb1 and PDSb2 were placed on the outside and inside of the glass shield of control room respectively. This glass shield would represent all personnel working in the operating theatre and marked as position B.
  Position B was 160 cm. above the floor.
  Interventions: Radiation: PDSb

INTERVENTIONS:
Radiation: PDSa — After an anesthesiologist administered a narcotic and an induction agent to a patient (total intravenous anesthesia, TIVA), an endoscopist commenced the procedure. A co-researcher turned on Pocket Radiation Dosimeter label as PDSa1 (outside lead apron),PDSa2 (inside lead apron).
  Arms: PDSa (Pocket radiation dosimeter a)
Radiation: PDSb — After an anesthesiologist administered a narcotic and an induction agent to a patient (total intravenous anesthesia, TIVA), an endoscopist commenced the procedure. A co-researcher turned on Pocket Radiation Dosimeter label as PDSb1 (outside lead apron), PDSb2 (inside lead apron).
  Arms: PDSb (Pocket radiation dosimeter b)

SUMMARY:
Radiation now becomes a dreadful effect as its outcomes are tremendous to be expected. As a result, anesthetists become an inevitable target to the radiation exposure since they have to monitor patients closely during the operation. Unfortunately, radiation may not have an immediate sequelae, but an accumulation of adverse effects.

These sequelae happen by means of direct exposure and reflection. The reflected rays is inversely proportional to the distance between the origin and the target. Practically, the radiation source can be protected by individual cover and glass shield.

Siriraj hospital is a tertiary, general university hospital with 2,200 beds. Annually, an Endoscopy centre has over 700 patients undergoing endoscopic retrograde cholangio pancreaticography (ERCP). Normally, fluoroscopy for pancreatic and biliary ducts visualisation is needed under anesthesia. Though the procedure is operated in a well-equipped, radiating-protection room; many medical personnel including 1-2 endoscopists, 2 scrub nurses, 1-2 anesthetists and 1 x-ray man, still have a chance of irradiation.

During ERCP, all medical personnel particularly anesthetists are rinsed by radiation from here and there. Though they always wear lead aprons and collar shields to protect themselves from the rays, they are normally in the position - less than 1 meter - close to the fluoroscopy.

Due to the advancement in technology, anesthetists can remotely monitor patients during the surgical procedure. This might cause a lesser effect of ray upon them. As a result, whether or not the positioning of anesthesia personnel relating to the distance of x-ray source would help to alleviate the effect of radiation exposure.

DETAILED DESCRIPTION:
This study has been approved by Siriraj IRB. Inclusion criteria were the patient who underwent ERCP procedure. Exclusion criteria were none. The project was terminated when 19 August 2016 A total of 222 cases was included without the need of informed consent.

At the Endoscopic unit A nurse anesthetist performed venous cannulation on the right forearm and transfused with 5% dextrose in half-strength normal saline. Then the patient was transferred to the ERCP theatre.

The patient was monitored with non-invasive blood pressure (NIBP), percutaneous arterial oxygen saturation (SpO2), and electrocardiogram (EKG) and administered with oxygen 3LPM via nasal cannula.

A co-researcher reset and prepared 4 pocket dosimeters (PDS) and labelled as PDSa1, PDSa2, PDSb1 and PDSb2.

The PDSa1 and PDSa2 were placed on the outside and inside of a lead shirt respectively. The shirt-covered box was close to an anesthetic machine. This box would represent anesthetic personnel on duty and marked as position A.

The PDSb1 and PDSb2 were placed on the outside and inside of the glass shield of control room respectively. This glass shield would represent all personnel working in the operating theatre and marked as position B.

Both position A and B were 160 cm. above the floor. After an anesthesiologist administered a narcotic and an induction agent to a patient (total intravenous anaesthesia, TIVA), an endoscopist commenced the procedure. A co-researcher turned on all PDS devices as soon as the surgeon started a fluoroscopy, and turned it off whenever the use of radiative source was over. When the study was completed, the PDA devices was kept in a solid and dry place. The lead apron was hanged in the specific area and covered by a bag.

The devices

A lead apron was 0.5 mm. and 0.25 mm. in thickness on the front and back (BT medical) respectively. A thyroid shield was 0.5 mm. in thickness. A paper box was 30x1510 cm. in dimension. A radiative dosimeter (Ludlum model 25-IS &25-IS-1 Personal Radiation Monitor, 501 Oak street, Sweetwater, Texas, USA) had characteristic details as follow:

Ludlum model 25-IS & Model 25-IS-1 Radiation detected Gamma (X ray) typically < 18 count per minute per milliroentgen/hr.

Beta response typically < 0.10 milliroentgen/hr Display range For 25-IS: 0.01 milliroentgen/hr to 10 sievert/hr For 25-IS-1: 0.01 millisievert/hr to 10 sievert/hr Size. 7.6 x5.4x1.7 cm (H x W x thickness) Weight. 158.6 g. Including batteries Linearity. Reading within 10% of true value within calibration range

Analysis of data Data were expressed as mean and standard deviation and analysed by using SPSS version 18.0. Categorical data were compared by using Chi-square test; while, the recorded data using dependent t-test. A p < 0.05 was considered statistically significant difference at 95% confidence interval.

ELIGIBILITY:
Inclusion Criteria:

* The patient who underwent ERCP

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 222 (Actual)
Dates: Start 2015-09; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Amount of radiative difference | up to 1 year
  The amount of radiative difference on the outside of the shirt-covered box and the glass shield as compared to the inside.

CONTACTS AND LOCATIONS:
Overall Officials: Department of Anesthesiology Siriraj Hospital, Study Director — Department of Anesthesia, Faculty of Medicine Siriraj Hospital, Mahidol University

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] ASGE Technology Committee; Pedrosa MC, Farraye FA, Shergill AK, Banerjee S, Desilets D, Diehl DL, Kaul V, Kwon RS, Mamula P, Rodriguez SA, Varadarajulu S, Song LM, Tierney WM. Minimizing occupational hazards in endoscopy: personal protective equipment, radiation safety, and ergonomics. Gastrointest Endosc. 2010 Aug;72(2):227-35. doi: 10.1016/j.gie.2010.01.071. Epub 2010 May 26. PMID 20537638
- [Background] Ismail S, Khan F, Sultan N, Naqvi M. Radiation exposure to anaesthetists during interventional radiology. Anaesthesia. 2010 Jan;65(1):54-60. doi: 10.1111/j.1365-2044.2009.06166.x. Epub 2009 Nov 17. PMID 19922509
- [Background] Miller PS, Braiterman LT, Ts'o PO. Effects of a trinucleotide ethyl phosphotriester, Gmp(Et)Gmp(Et)U, on mammalian cells in culture. Biochemistry. 1977 May 3;16(9):1988-96. doi: 10.1021/bi00628a036. PMID 557989
- [Background] Markou P. [Fetus radiation doses from nuclear medicine and radiology diagnostic procedures. Potential risks and radiation protection instructions]. Hell J Nucl Med. 2007 Jan-Apr;10(1):48-55. Greek, Modern. PMID 17450255
- [Background] Daas AY, Agha A, Pinkas H, Mamel J, Brady PG. ERCP in pregnancy: is it safe? Gastroenterol Hepatol (N Y). 2009 Dec;5(12):851-5. PMID 20567530